CLINICAL TRIAL: NCT00971529
Title: Phase 1 Study on Smoking Cessation Effect of Tea Filter
Brief Title: Smoking Cessation Effect of Tea Filter Through Inhibition of Nicotine Receptor
Status: Completed | Type: Observational
Sponsor: General Hospital of Beijing PLA Military Region (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Ran Tao/, Beijing Military Region General Hospital
Other Study IDs: zhaotaoliang123
Record Dates: First submitted 2009-08-20; First posted 2009-09-03 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Tobacco Cessation
Keywords: Smoking cessation; tea filter
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — CO
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- lifestyle: 70 volunteers were double-blinded, placebo-controlled and randomized into 2 groups (smoking with tea filters or regular filters).
- tea filter: The investigators then recruited 59 volunteers with longer smoking history and stronger desire for quitting smoking for smoking cessation test using the tea filter.

SUMMARY:
Cigarette smoking is the major risk factor for a series of life threatening diseases including cancer and heart attack, which causes millions of deaths each year worldwide. Many of the harmful effects of cigarette smoking can be reversed by quitting; however, due to the addictive nature of nicotine, quitting smoking is extremely difficult. Despite the efforts, currently available methods produce only modest smoking cessation rates with relapse. Previously, tea components were shown to protect effect against cigarette smoke-induced toxicity. Here the investigator reported an unprecedented smoking cessation effect of tea. Green tea was made into cigarette filters and tested for its smoking cessation effect in a double-blind clinical study. The tea filter could effectively achieve abstinence relapse using smoking process to quite smoking and easy to be used by smoker without any side effects and psychological obstacles. This work provides a new idea and innovative method to combat tobacco epidemic. Its implementation and popularization may make a great contribution towards to reducing the smoking-related diseases, and relieving the public health burden and pollution caused by cigarette smoking.

DETAILED DESCRIPTION:
Cigarette smoking has been linked to many life threatening diseases including heart diseases, cancer and chronic obstructive pulmonary disease. There are about 1.25 billion smokers in the world. Five million people die every year because of smoking-related diseases. This rate exceeds many other diseases combined. It is estimated that the global cost for smoking-related diseases is about $200 billion each year, posing one of the biggest public human health problems around the world. Many methods have been developed for smoking cessation by scientists and doctors worldwide. However, due to the addictive nature of nicotine, quitting smoking is extremely difficult. Despite all the efforts, currently available smoking cessation methods produce only modest successful rates with relapse. In addition, they are often not convenient and can lead to a wide variety of side effects. Therefore, the need of new idea for developing new smoking cessation techniques with better efficacy and fewer side effects is urgent.

Epidemiological evidences have shown that tea is adversely associated with cancer, hyperglycemia and other diseases. In addition, we have shown that tea components protect cells from cigarette smoke-induced toxicity. Recently, we have developed a new cigarette filter containing tea. While testing the filter for detoxification effects, we found that several subjects who were smokers decreased their cigarette consumption and subsequently abstained from cigarette smoking after using the tea filter for a period of time. Animal experiments revealed that a derivative tea component prevented nicotine addiction similar to nicotine acetylcholine receptor (nAChR) inhibitor. It significantly inhibited the nicotine-induced expression of alpha4,alpha7 and β2 subunits of nAChR and tyrosine hydroxylase and release of dopamine. This finding encouraged us to recruit more volunteers to test the smoking cessation effect of the tea filter.

One hundred healthy male cigarette smokers, aged 18 to 30 years, were screened and 30 of them were excluded based on the exclusion/inclusion criteria. 70 volunteers were double-blinded, placebo-controlled and randomized into 2 groups (smoking with tea filters or regular filters). Smoking history, including the nicotine dependence, was assessed at the screening visit. Exclusion criteria included treatment with an investigational drug within the previous month; major depression within the prior year; panic disorder, psychosis, or bipolar disorder; use of nicotine replacement therapy or other drugs within the previous 3 months; cardiovascular disease; clinically significant medical disease; drug or alcohol abuse or dependence within the past year; and use of tobacco products other than cigarette smoking within the previous month. Subjects received brief smoking cessation counseling (up to 10 minutes) at the baseline visit and at each visit afterwards. Self-reported smoking status since the last visit and exhaled carbon monoxide measurement were assessed at each weekly visit. Vital signs, weight, and adverse event information were collected at each visit. A physical examination was performed prior to randomization and at the final visit. Urine and blood were collected at screening, baseline, and at weeks 1, 2, 3, and 4 for biochemical analysis.

The average number of cigarettes consumed daily by one volunteer smoker before the clinic trial was calculated as control. The average number of cigarettes consumed daily by one volunteer after the clinic trial was calculated and the numbers were then used to calculate the averages number of cigarettes consumed daily by one smoker in a week and compared with control. Continuous abstinence was defined as self-report of no cigarette use during the specified time period confirmed by an exhaled carbon monoxide measurement of 10 ppm or lower. To be considered abstinent from smoking during the treatment period, subjects also had to report that they did not use any other nicotine-containing products. During the follow-up period, use of nicotine replacement therapy did not disqualify subjects from being considered abstinent. Subjects who withdrew or were lost to follow-up were assumed to be smokers for the remainder of the study. The exhaled carbon monoxide was detected by a carbon monoxidemeter (1209-1 CO, DWYER, USA). Nicotine and cotinine in urine was detected using HPLC (HITACH, Japan) as reported in the literature.

30 volunteers in control group and 22 volunteer male cigarette smokers who consumed on average approximately cigarettes per day, were randomly divided into 2 groups (double-blind, placebo-controlled); smoking with tea filters or with regular filters. After using the tea filter for 1 month, the average daily cigarette consumption decreased about 43% in the tea filter group. In contrast, no change in average daily cigarette consumption was detected in the control group using regular filters. The trial was discontinued for the control group and the tea filter group was followed for another month. After using the tea filter for 2 months.

We then recruited 59 volunteers with longer smoking history and stronger desire for quitting smoking for smoking cessation test using the tea filter. The subjects were followed for 5 month following the same protocol as described earlier.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male cigarette smokers, aged 18 to 65 years

Exclusion Criteria:

* Exclusion criteria included treatment with an investigational drug within the previous month
* Major depression within the prior year
* Panic disorder
* Psychosis
* Bipolar disorder
* Use of nicotine replacement therapy or other drugs within the previous 3 months
* Cardiovascular disease
* Clinically significant medical disease
* Drug or alcohol abuse or dependence within the past year
* Use of tobacco products other than cigarette smoking within the previous month.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 70 volunteers were double-blinded, placebo-controlled and randomized into 2 groups (smoking with tea filters or regular filters).
  The investigators then recruited 59 volunteers with longer smoking history and stronger desire for quitting smoking for smoking cessation test using the tea filter.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
number of cigarettes consumed daily by every volunteer smoker | 1-5 months

SECONDARY OUTCOMES:
exhaled carbon monoxide by the volunteers | in the evening

CONTACTS AND LOCATIONS:
Overall Officials: Ran Tao, MD, Study Director — Addiction Branch, Beijing Military Reneral Hospital
Locations (1):
- Ran Tao, Beijing, China